CLINICAL TRIAL: NCT05833711
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Froniglutide (PF1801) in Patients With Idiopathic Inflammatory Myopathy (IIM)
Brief Title: Study Evaluating Efficacy and Safety of Froniglutide (PF1801) in Patients With Idiopathic Inflammatory Myopathy
Acronym: FROG
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Immunoforge Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PF1801-CL-202
Record Dates: First submitted 2023-04-16; First posted 2023-04-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dermatomyositis; Polymyositis; Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Dermatomyositis; Polymyositis; Myositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Froniglutide 50 mg (Experimental): Froniglutide (PF1801) 50 mg will be administered subcutaneously once a week.
  Interventions: Drug: Froniglutide
- Froniglutide 70 mg (Experimental): Froniglutide (PF1801) 70 mg will be administered subcutaneously once a week.
  Interventions: Drug: Froniglutide
- Placebo (Placebo Comparator): Matching placebo will be administered subcutaneously once a week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Froniglutide — SC Weekly Injection
  Other Names: PF1801
  Arms: Froniglutide 50 mg; Froniglutide 70 mg
Drug: Placebo — SC Weekly Injection
  Arms: Placebo

SUMMARY:
This is a Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Froniglutide in Patients With Idiopathic Inflammatory Myopathy ("FROniGlutide Study")

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of IIM (DM or polymyositis [PM]) as per Bohan and Peter classification criteria
* MMT-8 ≤125 units and two out of the following CSM items, or MMT-8 >125 units and three out of the following CSM items, together with verifiable muscular weakness A. PGA VAS ≥2 cm B. SGA VAS ≥2 cm C. HAQ-DI ≥0.25 D. Extramuscular activity (MDAAT) ≥2 cm E. Increase in one or more muscle enzyme (CK, LDH, AST, ALT, aldolase) values (must be ≥1.3 × ULN)
* On treatment with standard of care (immunosuppressants and/or corticosteroids) for >12 weeks and on stable therapy for at least 4 weeks

Key Exclusion Criteria:

* Inclusion body myositis (IBM) or amyopathic DM
* Severe muscle damage (myositis damage index [MDI] >7/10 cm). Permanent deterioration caused by reasons other than PM/DM, or myositis with cardiac involvement
* Clinically significant renal/hepatic impairment
* Severe interstitial lung disease requiring supportive oxygen therapy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
IMACS-TIS Moderate Improvement at Week 24 | Week 24
  Proportion of subjects who achieve moderate improvement (≥40) from baseline in IMACS TIS at Week 24

SECONDARY OUTCOMES:
IMACS-TIS Minimal Improvement at Week 4, 8, 12, 16, 24 | Week 4, 8, 12, 16, 24
  Proportion of subjects who achieve minimal improvement (≥20) from baseline in IMACS TIS at Week 4, 8, 12, 16, and 24

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea